CLINICAL TRIAL: NCT05550987
Title: Assessment of the Effectiveness of the Use of Modern Technologies in the Rehabilitation of Patients With Neurological Diseases
Brief Title: The Use of Modern Technologies in Neurorehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Rzeszow (Other)
Collaborators: Donum Corde Rehabilitation Center (Unknown)
Responsible Party: Principal Investigator, Agnieszka Wiśniowska-Szurlej, PhD, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neurorehabilitation
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Neurorehabilitation; Nervous System Diseases; Biomedical Enhancement; Physical Activity
Keywords: Exercise Therapy; Neurological Rehabilitation,; Recovery of Function
MeSH Terms: conditions — Nervous System Diseases; Motor Activity | interventions — Rehabilitation; Control Groups

STUDY DESIGN:
Intervention Model Description: Random selection to two groups (study group and control group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Vibramoov Device (Experimental): Rehabilitation program with the use of mechanical vibration using the Vibramoov device and conventional physiotherapy
  Interventions: Other: Control Group
- Ekso GT exoskeleton Device (Experimental): Rehabilitation program with gait training using the Ekso GT exoskeleton and conventional physiotherapy
  Interventions: Other: Control Group
- RoboGait Device (Experimental): Rehabilitation program with the use of gait training with the use of a RoboGait stationary robot and conventional physiotherapy.
  Interventions: Other: Control Group
- ZEBRIS Device (Experimental): Rehabilitation program with the use of gait training with the use of the ZEBRIS treadmill and conventional physiotherapy
  Interventions: Other: Control Group
- PABLO Device (Experimental): Rehabilitation program with the use of upper limb function training with the use of the PABLO device and conventional physiotherapy
  Interventions: Other: Control Group
- Control Group (Experimental): Rehabilitation program with conventional physiotherapy
  Interventions: Other: Rehabilitation program with the use of mechanical vibration using the Vibramoov device and conventional physiotherapy; Other: Rehabilitation program with gait training using the Ekso GT exoskeleton and conventional physiotherapy; Other: Rehabilitation program with the use of gait training with the use of a RoboGait stationary robot and conventional physiotherapy.; Other: Rehabilitation program with the use of gait training with the use of the ZEBRIS treadmill and conventional physiotherapy; Other: Rehabilitation program with the use of upper limb function training with the use of the PABLO device and conventional physiotherapy

INTERVENTIONS:
Other: Rehabilitation program with the use of mechanical vibration using the Vibramoov device and conventional physiotherapy — The Vibramoov device (Techno Concept, France) will be used in the rehabilitation program. Before starting the training session, each subject will undergo a diagnosis in order to qualify for the use of Functional Proprioceptive Vibration. Before starting the therapy, pads are placed on the patient's body to fix the vibrating modules in the places to be treated (lower limbs, left upper limb or right upper limb). Then the vibrating modules are attached to the supports. The therapy carried out with the use of the Vibramoov device consists in the targeted and individualized stimulation of the nervous system, as in the course of natural movements of the upper or lower limbs with the use of visual biofeedback. Therapy with the use of the Vibramoov device will be carried out 4 times a week for 50 minutes a day. Additionally, individual physiotherapy (50 minutes) and upright standing (50 minutes) will be conducted 5 times a week.
  Arms: Control Group
Other: Rehabilitation program with gait training using the Ekso GT exoskeleton and conventional physiotherapy — The Ekso GT ™ exoskeleton (Ekso Bionics, Inc. Richmond, CA, USA) used in the rehabilitation program has been approved by the Food and Drug Administration (FDA). Before starting the training session, each subject will undergo a thorough diagnosis to individually adjust the bionic skeleton. After entering the patient's data into the device's software, the physiotherapist selects the optimal training parameters. As the patient progresses during the training unit, the therapist will update the exoskeleton settings on an ongoing basis, so that the training is best suited to the current capabilities of the subject. Therapy with the use of the exoskeleton device will be carried out 4 times a week for 50 minutes a day. Additionally, individual physiotherapy (50 minutes) and upright standing (50 minutes) will be conducted 5 times a week.
  Arms: Control Group
Other: Rehabilitation program with the use of gait training with the use of a RoboGait stationary robot and conventional physiotherapy. — The RoboGait stationary robot (Bama technologist, Turkey) will be used in the rehabilitation program. Before starting the training session, each subject will undergo detailed diagnostics in order to individually adjust the orthoses. The next step will be to put on a vest and inguinal straps on a wheelchair or standing, and then lift it up with the device, then attach it to the Robogait orthoses. After entering the patient's data into the software of the device, the physiotherapist selects the optimal training parameters. During the session, biofeedback is also displayed informing the patient and the therapist about the patient's activity level in the transfer phase and the support during walking for both lower limbs. Therapy with the use of the RoboGait device will be carried out 4 times a week for 50 minutes a day. Additionally, individual physiotherapy (50 minutes) and upright standing (50 minutes) will be conducted 5 times a week.
  Arms: Control Group
Other: Rehabilitation program with the use of gait training with the use of the ZEBRIS treadmill and conventional physiotherapy — The Zebris FDM-T treadmill will be used in the rehabilitation program for gait analysis. Before each session, patients will be equipped with a harness for safety reasons. The need for a handrail will be assessed prior to each session and patients will be encouraged to support their hands as little as possible. Before starting the training session, each subject will undergo a thorough diagnosis in order to individually adjust the training parameters. Therapy with the use of the Zebris FDM-T treadmill will be carried out 4 times a week for 50 minutes a day. Additionally, individual physiotherapy (50 minutes) and upright standing (50 minutes) will be conducted 5 times a week.
  Arms: Control Group
Other: Rehabilitation program with the use of upper limb function training with the use of the PABLO device and conventional physiotherapy — The Pablo (Tyromotion) device will be used in the rehabilitation program. Before the start of the training session, each subject will undergo detailed diagnostics assessing the range of mobility in the shoulder, radiocarpal (frontal and sagittal plane), elbow (sagittal plane), and explosive strength of the cylindrical, pinch and lateral and three-point grip. The Force Control Index will also be designated. The next stage will be training on the Pablo device using visual and auditory biofeedback. The physiotherapist selects the optimal training parameters (type of pad, type of game, level of the game). Each training session will be stored in the software and recorded in the patient's medical records. Therapy with the use of the Pablo device will be carried out 4 times a week for 50 minutes a day. Additionally, individual physiotherapy (50 minutes) and upright standing (50 minutes) will be conducted 5 times a week.
  Arms: Control Group
Other: Control Group — In control Group the rehabilitation program will be carried out for a period of 4 weeks. In each of the studied groups, the rehabilitation program will include conventional physiotherapy sessions performed 5 times a week, consisting of 50 minutes a day of individual physiotherapy and 50 minutes a day of standing upright.
  Arms: Ekso GT exoskeleton Device; PABLO Device; RoboGait Device; Vibramoov Device; ZEBRIS Device

SUMMARY:
Early conventional rehabilitation improves the functioning of patients with neurological diseases. However, recovery is not always satisfactory. These needs are met by the constantly developing modern technologies supporting the process of neurorehabilitation. The main goal of the research project is to evaluate the use of modern technologies in the rehabilitation of patients with neurological diseases (after stroke, craniocerebral trauma, spinal cord injury, cerebral palsy and multiple sclerosis). According to the research hypothesis, intensive rehabilitation with the use of modern technologies will improve the functional efficiency of patients with neurological diseases.

DETAILED DESCRIPTION:
Study participants will be recruited from the Donum Corde Rehabilitation Center. After meeting the inclusion criteria, the qualification for the use of modern technologies in the rehabilitation process will be performed. After a patient is enrolled in one of the five study programs, study participants will be randomly assigned to the study group and the control group. Randomization will be performed by a statistician, a member of the research team. After randomization, the rehabilitation program will be carried out for a period of 4 weeks. In each of the studied groups, the rehabilitation program will include therapy with the use of modern technologies, performed 4 times a week, 50 minutes a day, and conventional physiotherapy sessions performed 5 times a week, consisting of 50 minutes a day of individual physiotherapy and 50 minutes a day of standing upright. Exercises will be performed by qualified physiotherapists with at least 3 years of experience in working with neurological patients. Therapies with the use of modern technologies will be performed by certified physiotherapists after training and courses in the use of modern rehabilitation devices. The improvement process will take place from Monday to Friday for 4 weeks, under the supervision of the Scientific and Medical Research Supervisor and the care and consent of the ward doctor. After 4 weeks of exercise, examination II will be performed after rehabilitation is complete. The obtained results will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 to 75;
* Body height <190 cm;
* Body weight <100 kg;
* Normal cognitive status - AMTS> 6;
* Doctor's consent to participate in the rehabilitation process;
* Informed consent of the examined person to participate in the study;
* Coexistence of a neurological disorder: post-stroke condition; craniocerebral trauma; multiple sclerosis; cerebral palsy; total or partial spinal cord injury; other neurological conditions characterized by a gait problem or an inability to walk and impaired function of the upper limb.

Exclusion Criteria:

* Severe coexisting diseases (infections, cardiovascular diseases, heart and lung diseases);
* Fracture of the lower limbs in the last 2 years;
* Osteoporosis or densitometry t-score less than -2.5 SD;
* Neurogenic periarticular ossification of the lower limbs;
* Pressure ulcers or wounds in the lower limbs;
* Spasticity> 4 on the Ashwort scale;
* Pregnancy;
* Colostomy;
* Lower limb prostheses or arthroplasty;
* Significant limitations in the range of motion and pain (hip, knee and ankle joints) that make it difficult to move

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
An assessment of static and dynamic balance using Berg Balance Scale (BBS) | at baseline, immediately after treatment
  Assessment of static and dynamic balance based on 14 types of movement in the standing and sitting position of the patient. Each task of the test is scored using a four-point scale. A maximum score of 56 points is possible. Patients with a score below 20 pts indicate high risk of fall and the need of using wheelchairs.
An assessment of locomotor stages after Spinal Cord Injury using LOSSCI Scale | at baseline, immediately after treatment completion
  The LOSSCI is a five-stage scale result of applying and adapting to spinal cord injury the original Vojta's 10 specific locomotor stages. Each LOSSCI stage should be evaluated in ascending order and the grading is determined by the highest stage the person can accomplish: orienting to and touching or grasping an object in supine position, trunk uprighting in prone position, creeping, crawling or walking support for the upper limbs, independent bipedal locomotion. The person's highest stage is reached when at least one item in a stage is achieved.
An assessment of trunk movement using The Trunk Control Test for Motor Impairment After Stroke (TCT) | at baseline, immediately after treatment completion
  The TCT examines four axial movements: rolling from a supine position to the weak side and to the strong side, sitting up from a lying-down position, and sitting in a balanced position on the edge of the bed with feet off the ground for 30 seconds. The scoring is as follows: 0, unable to perform movement without assistance; 12, able to perform movement but in an abnormal manner; and 25, able to complete movement normally. The TCT score is the sum of the scores obtained on the four tests (range, 0 to 100).
An assessment of fall risk using Timed Up and Go Test (TUG) | at baseline, immediately after treatment completion
  Measurement of the time in seconds for a person to rise from sitting from a standard arm chair, walk 3 meters, turn, walk back to the chair, and sit down.
An assessment of motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale | at baseline, immediately after treatment completion
  Fugl-Meyer Motor Assessment Scale for Upper Extremity is a comprehensive tool enabling measurement of motor function; it comprises 33 motor tasks, designed to assess general movements, precision movements, grip, coordination and speed. It is also possible to perform H subgroup tests - assessing superficial and deep sensibility, and J subgroup tests - for range of passive motion and pain induced by such movements. Individual tasks are assessed on a scale 0-2 0 - impossible task. The higher the score, the better.

SECONDARY OUTCOMES:
An assessment of muscle tone using modified Tardieu Scale | at baseline, immediately after treatment completion
  The scale takes into account the tension depending on the bending speed of the limb. It includes an assessment of the extent of passive motion when a muscle is stretched at a very slow pace, an assessment of the quality of the muscle's response during rapid stretching, and a measurement of the angle at which the muscle first responds to overactive stretching.
An assessment of the parameters describing the center of pressure of the feet for measurements with eyes open and closed carried out on the stabilometric platform ALFA | at baseline, immediately after treatment completion
  The balance will be conducted using the Alfa platform. The board platform will be set up in parallel, 2 m from the walls of the room, where a tag will be placed to focus vision with open eyes during the trials. The measuring device will be calibrated before each test. The study will consist of two 30-s trials performed with open and closed eyes. The participant will be asked to conduct the test without shoes, in a relaxed standing position, with arms down by the sides.
An assessment of strength and quality of grips carried out on the Pablo | at baseline, immediately after treatment completion
  Assessment of the strength of a cylindrical grip and extension as well as grips: pincer, lateral, two-point, three-point measured in kilograms and the force control index (0-100 points). The force control index is determined on the basis of: force reaction time, release time, force value exceeding, bending and extension time control.
Analysis of gait spatiotemporal parameters carried out on Zebris | at baseline, immediately after treatment completion
  The Zebris FDM-T is fitted with an electronic mat of 10,240 miniature force sensors, each approximately 0.85 × 0.85 cm embedded underneath the belt. The treadmill's contact surface measures 150 × 50 cm and its speed can be adjusted from 0.2 to 22 km/h, at intervals of 0.1 km/h. When the subject will stands/walks on the treadmill, the force will be exerted by his feet (the so-called reactive-normal force) and recorded by the sensors at a sampling rate of 120 Hz. Dedicated software will be integrated the force signals and provides 2D/3D graphic representation of major spatiotemporal parameters.
Analysis of isometric muscle strength carried out on RoboGait | at baseline, immediately after treatment completion
  Based on the gait analysis carried out with the RoboGait, the isometric muscle strength will be obtained.
Analysis of gait carried out on Ekso Skeleton | at baseline, immediately after treatment completion
  The EksoGT powered robotic exoskeleton will be used to provide the experimental intervention for this study. The number of steps during training will be assessed.
An assessment of manual skills using Box and Blocks Test | at baseline, immediately after treatment completion
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds
An assessment of handgrip function using Franchay scale | at baseline, immediately after treatment completion
  The scale consists of 7 tasks (pass/fail grading); the patient is awarded 1 point for each activity performed successfully, or 0 points for a failure to perform. The maximum score of seven points may be achieved for the performance of the tasks. Higher score corresponds to better manual skills. The scale measures the proximal control of the upper limb and the manual skills
An assessment of ability to perform basic activities of daily living using Barthel Index | at baseline, immediately after treatment completion
  Barthel Index is a scale for ADL (Activities of Daily Living) measurement, with lower scores indicating greater dependency in ADL. The score value ranges between 0 and 100 points. The assessment of the total score is as follows: 0-20 completely dependent; 21-61 almost completely dependent; 62-85 dependent; 91-100 - independent
An assessment of body composition using subjected to bioelectrical impedancy analysis - Tanita 780 | at baseline, immediately after treatment completion
  The TANITA is an 8-contact electrode system capable of acquiring segmental body composition analysis without the need for gel electrodes. Measurements using the TAN segmental body composition analyzer were recorded following a standardized 10-min standing period to minimize acute shifts in fluid distribution. Subject details were entered into the TAN, including information on clothing weight, gender, age, and height. When prompted, subjects stepped onto the footpads and grasped the handles. Analysis took approximately 10 sec during which time the subjects remained still and relaxed. Measurements were recorded in the standard mode.
An assessment of quality of life using The World Health Organization quality of life (WHOQOL) - BREF | at baseline, immediately after treatment completion
  The WHOQOL-Bref questionnaire was used to assess the quality of life, which allows to obtain a profile of quality of life on the basis of the analysis of the last 14 days in four domains: physical, psychological, social and environmental. Answers to the questions asked are classified in a five-point scale, and the interpretation of the obtained results has a positive direction. This means that the greater the number of points scored in each of the assessed domains, the better the quality of life of the subject.
An assessment of level of disability using The World Health Organization Disability Assessment Schedule (WHODAS 2.0) | at baseline, immediately after treatment completion
  The questionnaire enables the assessment of the functioning of people in the last 30 days in six domains of life: understanding and communicating, getting around, self-care, getting along with people, life activities and participation in society. Answers to the questions were classified in a five-point scale in which, along with the increase in the score obtained, the severity of the problem increases (no problem - 1 point, extremely big problem - 5 points). After summing up the results obtained in each of six domains and converting them to the 0-100 point range, it is also possible to assess the overall disability level, in which 0 points means no disability and 100 points - total disability
An assessment of Lung Capacity assessment using a peak expiratory flow (PEV) measurement | at baseline, immediately after treatment completion
  Lung Capacity was measured based on peak expiratory flow (PEF) and forced expiratory volume in 1 second (FEV1) using Peak flow meter (Peak Flow Meter Microlife PF 100, measuring range: 50-900 l/min and FEV1 0,01-9,99 l). Participants take a deep breath and blow air into the meter as fast as they can. For PEF and FEV1, at least three measurements were performed until the best values was selected
An assessment of walking speed using the 10 meter walk test (10MTW) | at baseline, immediately after treatment completion
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.

OTHER OUTCOMES:
An assessment of cognitive state using The abbreviated mental test score (AMTS) | at baseline, immediately after treatment completion
  The Abbreviated Mental Test Score (AMTS) is a tool designed for the assessment of cognitive functions, such as episodic memory, semantic memory and working memory, to screen for potential problems in cognitive functioning. AMTS is a 10-item questionnaire comprising questions and simple tasks for the patient. It takes only several minutes to perform, is simple, and no professional knowledge or equipment are needed.
An assessment of anxiety and depression using Hospital Anxiety and Depression Scale (HADS) | at baseline, immediately after treatment completion
  The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately. Cut-off scores are available for quantification, for both scales, scores of less than 7 indicate non-cases.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Wiśniowska-Szurlej, Principal Investigator — University of Rzeszow

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available from the corresponding author, upon reasonable request.